CLINICAL TRIAL: NCT05308407
Title: POWER UP: Participating Online While Exercising to Recover Using Play
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: <75% participation
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-0887; NCI-2022-02423 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2022-03-15; First posted 2022-04-04 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Exercise; Central Nervous System Tumors; Tumors
MeSH Terms: conditions — Motor Activity; Central Nervous System Neoplasms; Neoplasms | interventions — Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aim 1. Focus Groups (Other): Healthcare providers (n=16-24 participants in 4 focus groups) from MD Anderson Cancer Center (MDACC).
  AYAs with primary benign or malignant central nervous system tumors (n=16-24 participants in 4 focus groups) treated at MDACC.
  Interventions: Other: Focus Groups
- Aim 2. Pilot randomized controlled trial: (Other): AYAs with primary benign or malignant central nervous system tumors (n=80 patients approached, with n= 40 participants consented and randomized to the intervention (n=20) or usual care control group (n=20)) treated at MDACC, any gender and race, who are ≤1-year post-surgery for a central nervous system tumor.
  Interventions: Other: Pilot randomized controlled trial

INTERVENTIONS:
Other: Focus Groups — No intervention involved in this phase of the study
  Arms: Aim 1. Focus Groups
Other: Pilot randomized controlled trial — The intervention is a virtually delivered, 12 weekly group-based active video game-centered lifestyle physical activity intervention (POWER UP) targeting affect to improve function and quality of life in insufficiently active AYAs with central nervous system tumors.
  Arms: Aim 2. Pilot randomized controlled trial:

SUMMARY:
We will conduct a two-phase study. The first phase is to adapt and develop an active video game (AVG)-centered lifestyle physical activity (PA) intervention (POWER UP) for adolescents and young adults (AYA) with central nervous system tumors. The second phase is to test the feasibility and preliminary efficacy of a 12-week virtually delivered, group-based active video game-centered lifestyle physical activity intervention on function and quality of life in AYAs (aged 15-39) who are ≤1-year post-surgery for a central nervous system tumor. This population is at very high-risk for steep functional decline.

DETAILED DESCRIPTION:
Objective:

To develop (Aim 1) and test (Aim2, Primary Objective) the feasibility and acceptability of a virtually delivered, group-based active video game-centered lifestyle physical activity intervention targeting affect to improve function and quality of life in insufficiently active AYAs with central nervous system tumors. Also, (Aim 2, Secondary Objective) in a pilot randomized trial, compare the physical function, quality of live, and physical activity level between intervention and control groups.

Primary: Feasibility and acceptability of the POWER UP intervention and assessments.

Secondary: Physical function, quality of life (QOL), symptoms, and PA levels as measured at the 12- and 24-week follow ups

. Other endpoints relevant to the primary and secondary objectives: BMI status, dietary intake, Fitbit data (days worn and steps), exercise motivation, basic psychological needs at the 12- and 24-week follow-ups

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in Aim 1 of this study, an individual must meet all of the following criteria:

Round 1 focus groups:

1. Oncologists who are caring for AYA cancer survivors or
2. Survivorship care providers who actively engage with AYA cancer survivors

Round 2 focus groups:

1. AYA cancer survivors age 15-39 years old
2. Self-reported diagnosis of a primary benign or malignant CNS tumor or confirmed diagnosis of primary benign or malignant CNS tumor radiographically or pathologically when available
3. ≤1-year post surgery and can have other tumor-directed treatment (e.g., radiation and/or chemotherapy)
4. Participants and/or guardians are willing and able to provide informed consent
5. Able to speak, read, and understand English
6. Daily access to the web
7. Can receive physical therapy because this is part of the standard of care

In order to be eligible to participate in Aim 2 of this study, an individual must meet all of the following criteria:

1. Age 15-39 years old
2. Self-reported diagnosis of a primary benign or malignant CNS tumor or confirmed diagnosis of primary benign or malignant CNS tumor radiographically or pathologically when available
3. ≤1-year post surgery and can have other tumor-directed treatment (e.g., radiation and/or chemotherapy)
4. Participant is insufficiently active (reports less than 150 minutes of planned moderate-vigorous intensity activity per week in the prior week)
5. Able to speak, read, and understand English
6. Daily access to the web
7. Approval to participate from the oncology care team
8. Participants and/or guardians are willing and able to provide informed consent
9. Able to move arms and legs as well as ambulate safely with and without a gait aid
10. Available space on the smartphone to download required apps
11. Can receive physical therapy because this is part of the standard of care
12. Participants and/or guardians are willing and able to provide informed consent for protocol PA18-0130 (Pediatric Energy Balance Data Repository Study), companion protocol for the Fitbit application/assessment.

Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in Aim 1 of this study:

Round 1 Focus Groups:

1. Do not have access to the internet

Round 2 Focus Groups:

1. Another member of the household is a participant or staff member on this trial
2. Do not have access to the internet
3. In foster care or is incarcerated
4. Cognitive and/or major sensory deficits that would impede the completion of research activities and assessments as deemed by the clinical team.
5. Self-reported diagnosis of a metastatic CNS tumor or confirmed diagnosis of a metastatic CNS tumor radiographically or pathologically when available

An individual who meets any of the following criteria will be excluded from participation in Aim 2 of this study:

1. Currently pregnant
2. Currently have dementia
3. Plans to travel for more than 2 weeks at a time during the study period where the participant is not able to sign in to join the videoconferencing sessions
4. Clinical judgment by the oncology care team concerning safety based on the Physical Activity Readiness Questionnaire for Everyone (2020 PAR-Q+)
5. Cognitive and/or major sensory deficits that would impede the completion of research activities and assessments as deemed by the clinical team.
6. Self-reported diagnosis of a metastatic CNS tumor or confirmed diagnosis of a metastatic CNS tumor radiographically or pathologically when available
7. Currently participating in an organized commercial or research-based exercise program
8. Another member of the household is a participant or staff member on this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Quality of Life Questionnaire | through study completion, an average of 1 year
  PROMIS 29 includes the following domains
  * Physical Function (5=without any difficulty, 1=unable to do)
  * Anxiety (5=always, 1=never)
  * Depression (5=always, 1=never)
  * Fatigue (5=very much, 1=not at all)
  * Sleep Disturbance (5=very poor, 1=very good)
  * Ability to participate in Social Roles and Activities(5=never, 1=always)
  * Pain Interference (5=very much, 1=not at all)
  * Pain Intensity (10=worst pain imaginable, 0=no pain)

CONTACTS AND LOCATIONS:
Overall Officials: Keri L Schadler, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2025-04-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT05308407/ICF_000.pdf